CLINICAL TRIAL: NCT02558504
Title: Clinical and Medico-economic Evaluation of Radiofrequency Ablation Versus Oesophagectomy in the Treatment of High Grade Dysplasia in Barrett's Oesophagus
Brief Title: Radiofrequency in the Treatment of Barrett's Oesophagus
Acronym: HARMONI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-687
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Neoplasm
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oesophagectomy (Active Comparator): While surgical reference technique for invasive cancer of the lower esophagus is the technique according to Lewis Santy, there is no consensus on the technique and surgical approaches lack of specific work in the particular case of superficial lesions . The centers will have the choice of using the technique according to Lewis Santy with gastric plasty or technique of esophagectomy without thoracotomy with lower mediastinal dissection. In the absence of consensus to date available, abdominal surgery time will be by laparotomy or laparoscopy (laparoscopic assisted technique called). In both cases, an exploratory laparoscopy for diagnostic purposes is realized to remove an extension of the disease that would indicate against-resection with curative intent. For surgery, patients will be put under antisecretory therapy proton-pump inhibitor; this at least throughout the duration of the study.
  Interventions: Procedure: Oesophagectomy
- Radiofrequency ablation (Experimental): The equipment processing is:
  * The radiofrequency generator,
  * The radiofrequency balloon 360,
  * the radiofrequency probe 90.
  The radiofrequency treatment should be carried out according to the following protocol:
  * The radiofrequency treatment is done within 2 months following the last endoscopic assessment.
  * The maximum number of sessions is 4, including 2 maximum with 360 Halo probe.
  * Endoscopy is performed under general anesthesia.
  * The removal must begin at the top 1cm above the upper pole of the lesion and must end 1cm below the lower pole of the lesion.
  * The patient is left fasting until morning. In case of chest pain, the patient may receive analgesics.
  * During the time of treatment, the patient must follow an antisecretory therapy pump inhibitor with dual proton dose orally. The patient should avoid taking aspirin or nonsteroidal anti-inflammatory drugs during the 10 days following each session.
  Interventions: Device: Radiofrequency ablation

INTERVENTIONS:
Procedure: Oesophagectomy
  Arms: Oesophagectomy
Device: Radiofrequency ablation
  Other Names: esophageal radiofrequency
  Arms: Radiofrequency ablation

SUMMARY:
First intent treatment for superficial circular esophageal neoplasm is surgical resection. Endoscopic mucosal resection is not recommended due to the high rate of subsequent esophageal stenosis (higher than 80%).

Surgical limits are related to a high level of morbidity due, in particular, to respiratory complications or infections that require prolonged hospitalisations, and by significant rate of mortality (from 2 to 5 %). As an alternative to the surgical treatment, an innovative technique to remove esophageal circular preneoplastic and neoplastic lesions has been developed: it consists to ablate the mucosa by means of a balloon of a fixed diameter which incorporates approximately 100 electrodes on its surface that emit radiofrequency waves (HALO® Radiofrequency Ablation Technology System). By varying the strength and the duration of the electrical impulses, it is possible to obtain a homogenous and controlled destruction of the tissue of the whole mucosa, leaving no remaining pre-neoplastic or neoplastic elements underneath. The technique will be used for high grade glandular epithelial neoplasia, Vienna 4-1 or 4-2, developed on a mucosa at risk, i.e. the Barrett's oesophagus, occupying more than half of the circumference of the esophagus and that requires surgical treatment. The expected benefit for the patient is linked to the reduced invasiveness of the technique in comparison to the surgery

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years,
* General Condition WHO 0, 1 or 2,
* ASA Class I and II, eligible for endoscopic or surgical treatment with curative intent,
* Histological diagnosis of high grade glandular epithelial neoplasia (Vienna 4-1 to 4-46), possibly multifocal or stage 0 (Tis, N0, M0),
* Endoscopic and histological confirmed diagnosis of intestinal metaplasia,
* Histological diagnosis confirmed by two endoscopies with biopsies and two pathological readings; biopsies should be carried out according to the protocol of the SFED (four-quadrant biopsies every cm) with at least once acetic acid for staining. Operators describe Barrett's esophagus using he SFED planimetric model. The final exam will be no more than two months before the date of treatment and should have been achieved in investigator establishment,
* Extension height of Barrett's esophagus upstream of the upper part of the gastric folds or palisade vessels:

  * Minimum 1 cm,
  * Maximum 12 cm.
* In case of previous treatment by mucosal resection or submucosal dissection (DSM) for severe dysplasia or microinvasive carcinoma:

  * the resected lesion must have been well differentiated and confined to the muscular mucosa (m3 maximum) on histological analysis,
  * resection should be more than two months,
  * resection must have been macroscopically complete laterally,
  * resection must have been histologically complete in depth,
  * resection must have been histologically complete laterally with regard to the microinvasive cancer, that is to say with a clear margin of safety (margin may be high-grade dysplasia provided that the latter has not macroscopic translation),
  * At least one endoscopic and histologic follow-up should be conducted with dye in a period of less than two months before the date of treatment, and at the investigator establishment.
* Patient may take an inhibitor of proton pump equivalent to 2 times 40 mg of esomeprazole,
* No mediastinal or celiac, or suspected metastatic lymph nodes by EUS,
* Affiliation to a social security system or similar,
* Lack of participation in another clinical study,
* Informed consent signed.

Exclusion Criteria:

* - Aged under 18,
* Lack of informed consent signed,
* Radiofrequency treatment history,
* on going neoplastic history with a short prognosis,
* Concomitant participation in another clinical study
* Contraindication to general anesthesia,
* Patient with an esophageal location of scleroderma
* Presence of a cardiac pacemaker or stimulator
* Pregnant women or likely to be in the absence of effective contraception,
* Esophageal stenosis preventing the passage of an endoscope,
* Histology other than glandular neoplasia,
* History of or current history of esophageal cancer invading the submucosal layer of the esophagus or more,
* Surgical treatment history (except anti-reflux treatment) or esophageal radiotherapy,
* previous esophageal treatment by another method ablation: photodynamic therapy, argon plasma coagulation, laser, ....
* Esophageal varices observed in endoscopy,
* Coagulopathy or taking anticoagulants responsible an INR> 1.3 or a platelet count <75,000 per microL,
* Life expectancy of less than 3 years, due to intercurrent disease, especially neoplastic,
* Severe Medical pathology:

  * Liver cirrhosis (Child-Pugh all stages)
  * Respiratory failure:

VEMS (Maximum Expiratory Volume Second) <1L / min

PaO2 <60 mmHg

PaCO2> 45 mmHg

* Renal failure (Cl Cr < 60 mL /min /1,73m²),
* Heart attack within the last six months or progressive coronary artery disease,
* Severe distal arteriopathie > stage II of Leriche and Fontaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-01-07 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
complete histological eradication of the high grade glandular epithelial neoplasia | 12 months after the end of treatment
  The rate of success of the technique, success being defined as the complete histological eradication of the high grade glandular epithelial neoplasia without death attributable to the procedure. The relation of a death to the procedure will be determined by a committee of experts consisting of 3 surgeons or 3 hepatogastroenterologists depending on the arm, who do not participate to the study.

SECONDARY OUTCOMES:
Rate of complete histological eradication of Barret's oesophagus | 12 months after the end of treatment
Rate of mortality all causes merged | 12 months after the end of treatment
Rate of mortality attributable to the procedure | 30 days after end of the treatment
Percentage of patients with severe adverse reaction and minor adverse reactions linked to the procedure used, described by anatomical site | 30 days and 12 months after end of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Hépatogastroentérologie, Pavillon H, Hôpital Edouard Herriot, Lyon, France

REFERENCES:
- [Background] Barret M, Pioche M, Terris B, Ponchon T, Cholet F, Zerbib F, Chabrun E, Le Rhun M, Coron E, Giovannini M, Caillol F, Laugier R, Jacques J, Legros R, Boustiere C, Rahmi G, Metivier-Cesbron E, Vanbiervliet G, Bauret P, Escourrou J, Branche J, Jilet L, Abdoul H, Kaddour N, Leblanc S, Bensoussan M, Prat F, Chaussade S. Endoscopic radiofrequency ablation or surveillance in patients with Barrett's oesophagus with confirmed low-grade dysplasia: a multicentre randomised trial. Gut. 2021 Jun;70(6):1014-1022. doi: 10.1136/gutjnl-2020-322082. Epub 2021 Mar 8. PMID 33685969